CLINICAL TRIAL: NCT01983501
Title: A Phase 1b, Open-label Study to Assess the Safety and Tolerability of Tucatinib (ONT-380) Combined With Ado-trastuzumab Emtansine (Trastuzumab Emtansine; T-DM1)
Brief Title: A Study of Tucatinib (ONT-380) Combined With Ado-trastuzumab Emtansine (T-DM1) in Patients With HER2+ Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONT-380-004
Record Dates: First submitted 2013-10-28; First posted 2013-11-14 (Estimated); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: HER2 Positive Breast Cancers
Keywords: ONT-380; T-DM1; Kadcyla; Breast cancer; ARRY-380; Tucatinib
MeSH Terms: conditions — Breast Neoplasms | interventions — tucatinib; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tucatinib (ONT-380) in combination with T-DM1 (Experimental)
  Interventions: Drug: Tucatinib (ONT-380); Drug: T-DM1

INTERVENTIONS:
Drug: Tucatinib (ONT-380) — Given twice per day, orally
Drug: T-DM1 — Given intravenously once every 21 days
  Other Names: Kadcyla

SUMMARY:
The purpose of this study is to determine the maximal tolerated dose (MTD) or recommended dose (RD) and to assess the safety and tolerability of tucatinib (ONT-380) combined with ado-trastuzumab emtansine (T-DM1) in patients with HER2+ breast cancer.

DETAILED DESCRIPTION:
This is a Phase 1b, open-label study of tucatinib (ONT-380) given in combination with ado-trastuzumab emtansine (T-DM1) to patients with HER2+ breast cancer.

This study will use a 3+3 dose escalation design to evaluate up to four dose levels of tucatinib ONT-380 in order to identify the maximal tolerated dose/recommended dose (MTD/RD) of tucatinib (ONT-380) in combination with T-DM1. T-DM1 will be administered intravenously on day 1 of each cycle (except cycle 1, when it will be administered on day 2 to allow for PK assessments of tucatinib (ONT-380) alone).Tucatinib (ONT-380) will be administered orally, twice per day on days 1-21 of each cycle.

There will be 3-6 evaluable patients enrolled in each cohort in the dose escalation phase, unless that dose is found to be intolerable prior to completion of enrollment. At least 6 evaluable patients are to be treated at a dose level in order for an MTD/RD to be declared. Once an MTD/RD is declared, an additional 24 evaluable patients will be in enrolled in a MTD/RD expansion cohort for a total of 30 evaluable patients to be treated at the MTD/RD.

In addition to the MTD/RD expansion cohort, an optional additional cohort of up to 15 evaluable patients with either untreated, asymptomatic CNS metastases not needing immediate local therapy or progressive CNS metastasis following local therapy may also be enrolled and treated at the MTD/RD. Up to 63 evaluable patients may be treated in this study.

ELIGIBILITY:
Inclusion Criteria:

* HER2+ metastatic breast cancer, documented as HER2+ by FISH and/or 3+ staining by immunohistochemistry.
* History of prior therapy with trastuzumab and a taxane, separately or in combination. For patients in dose escalation and MTD expansion cohorts, prior therapy with trastuzumab and a taxane must have been for metastatic disease. For patients in CNS disease expansion cohorts, trastuzumab and taxane (together or separately) may have been given at any time prior to study enrollment as part of neoadjuvant therapy, adjuvant therapy, or therapy for metastatic disease.
* If female and of child-bearing potential, has negative pregnancy test within 14 days prior to treatment.
* If a sexually active male or a sexually active female of child-bearing potential, agrees to use dual (two concurrent) forms of medically accepted contraception from the time of consent until 6 months after the last dose of either tucatinib (ONT-380) or T-DM1, whichever is longer.
* Signed an informed consent document that has been approved by an institutional review board or independent ethics committee (IRB/IEC).
* Must have target or non-target lesions as per RECIST 1.1.
* All toxicity related to prior cancer therapies must have resolved to ≤ Grade 1, with the following exceptions: alopecia; neuropathy, which must have to resolved to ≤ Grade 2; and congestive heart failure (CHF), which must have been ≤ Grade 1 in severity and must have resolved completely.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at screening.
* In the opinion of the Investigator, life expectancy > 6 months.
* Adequate hematologic function as defined by:

  * Hemoglobin ≥ 9 g/dL
  * Absolute neutrophil count (ANC) ≥ 1000 cells/µL
  * Platelets ≥ 100,000/µL
* Adequate hepatic function as defined by the following:

  * Total bilirubin ≤ 1.5 X upper limit of normal (ULN)
  * Transaminases (aspartate aminotransferase/serum glutamic oxaloacetic transaminase [AST/SGOT] and alanine aminotransferase/serum glutamic pyruvic transaminase [ALT/SGPT]) ≤ 1.5 X ULN (< 2.5 X ULN if liver metastases are present)
* INR and aPTT < 1.5 X ULN unless on medication known to alter INR and aPTT.
* Calculated creatinine clearance ≥ 60 mL/min.
* Left ventricular ejection fraction (LVEF) must be within institutional limits of normal as assessed by echocardiogram or multigated acquisition scan (MUGA) documented within 4 weeks prior to first dose of study drug.

Exclusion Criteria:

* Medical, social, or psychosocial factors that, in the opinion of the Investigator, could impact safety or compliance with study procedures.
* Patient is breastfeeding.
* Patient was treated with any experimental agent within 14 days or five half-lives of study treatment, whichever is greater.
* Patient was treated with trastuzumab or other antibody based therapy within three weeks of starting study treatment or with chemotherapy or hormonal cancer therapy within two weeks of starting study treatment.
* Patient had prior exposure to a cumulative dose of doxorubicin that exceeded 360 mg/m2 or its equivalent.
* Previous treatment with T-DM1 at any time; or previous treatment with any small molecule HER2 inhibitors including (but not limited to) lapatinib, neratinib, or afatinib within the last 4 weeks prior to initiation of study therapy.
* CNS disease:

  * Patients with leptomeningeal disease are excluded
  * Dose escalation and MTD/RP2D expansion cohort: Patients with symptomatic CNS metastases are excluded. Patients with treated CNS metastases or untreated asymptomatic CNS metastases not requiring immediate local therapy may be eligible. Enrollment of patients with metastases must be approved by the study medical monitor.
  * Optional CNS disease expansion cohort: Patients with asymptomatic untreated CNS metastases not needing immediate local therapy or patients with progressive CNS disease following local therapy may be eligible with medical monitor approval.
* History of allergic reactions to compounds of similar chemical or biological composition to T-DM1 or tucatinib (ONT-380), except for a history of Grade 1 or Grade 2 Infusion Related Reaction to trastuzumab which has been successfully managed.
* Patients with uncorrectable electrolyte abnormalities.
* Known to be HIV positive. HIV testing is not required for those patients who are not known to be positive.
* Known carrier of Hepatitis B and / or Hepatitis C (whether active disease or not).
* Known liver disease, autoimmune hepatitis, or sclerosing cholangitis.
* Inability to swallow pills or any significant gastrointestinal diseases, which would preclude adequate absorption of oral medications.
* Use of a strong CYP3A4 inhibitor within three elimination half-lives of the inhibitor prior to the start of study treatment.
* Use of a strong CYP2C8 inducer or inhibitor within three elimination half-lives of the inducer or inhibitor prior to the start of study treatment.
* Radiotherapy within 14 days of study treatment; patient must have recovered from acute effects of radiotherapy to baseline.
* Known impaired cardiac function or clinically significant cardiac disease such as ventricular arrhythmia requiring therapy, congestive heart failure and uncontrolled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure > 100 mmHg on antihypertensive medications).
* Myocardial infarction or unstable angina within 6 months prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-02-28 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2020-09-03 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 12 months

SECONDARY OUTCOMES:
Incidence of clinical lab abnormalities | 12 months
Frequency of dose reductions in tucatinib | 12 months
Frequency of dose reductions in T-DM1 | 12 months
Objective response rate (ORR) | 12 months
Duration of response | 12 months
Disease control rate (DCR) | 12 months
  Defined as best response of complete response (CR), partial response (PR), or stable disease (SD)
Clinical benefit rate (CBR) | 12 months
  Defined as SD for ≥6 months, PR, or CR
Progression-free survival (PFS) | Up to approximately 6 years

CONTACTS AND LOCATIONS:
Overall Officials: JoAl Mayor, PharmD, BCOP, Study Director — Seagen Inc.; Corinna Palanca-Wessels, MD, PhD, Study Director — Seagen Inc.
Locations (11):
- United States (7):
  - University of Alabama, Birmingham, Alabama
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Kansas, Kansas City, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Providence Cancer Center, Portland, Oregon
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Northwest Medical Specialties, Tacoma, Washington
- Canada (4):
  - London Health Sciences Centre, London, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Hospital de la Cite-de-la-Sante, Laval, Quebec
  - Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Zhang D, Taylor A, Zhao JJ, Endres CJ, Topletz-Erickson A. Population Pharmacokinetic Analysis of Tucatinib in Healthy Participants and Patients with Breast Cancer or Colorectal Cancer. Clin Pharmacokinet. 2024 Oct;63(10):1477-1487. doi: 10.1007/s40262-024-01412-0. Epub 2024 Oct 5. PMID 39368039
- [Derived] Borges VF, Ferrario C, Aucoin N, Falkson C, Khan Q, Krop I, Welch S, Conlin A, Chaves J, Bedard PL, Chamberlain M, Gray T, Vo A, Hamilton E. Tucatinib Combined With Ado-Trastuzumab Emtansine in Advanced ERBB2/HER2-Positive Metastatic Breast Cancer: A Phase 1b Clinical Trial. JAMA Oncol. 2018 Sep 1;4(9):1214-1220. doi: 10.1001/jamaoncol.2018.1812. PMID 29955792